CLINICAL TRIAL: NCT02979054
Title: Performance and Safety Assessment of T4020 in Managing Corneal Epithelial Defect Following Epi-off Accelerated Crosslinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: LT4020-302
Record Dates: First submitted 2016-11-09; First posted 2016-12-01 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- T4020 (Experimental): 1 drop every other day during 5 days
  Interventions: Device: T4020
- Saline solution (Placebo Comparator): 1 drop every other day during 5 days
  Interventions: Device: Placebo

INTERVENTIONS:
Device: T4020
  Arms: T4020
Device: Placebo
  Arms: Saline solution

SUMMARY:
The purpose of this study is to assess the performance and safety of T4020 versus saline solution.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with progressive keratoconus
* Patients who signed and dated informed consent

Exclusion Criteria:

* Patient under 18 years
* History within 1 month or any active ocular infection, ocular injury, and associated corneal ulceration and abscess
* Corneal thickness< 400µm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Hospital, Varna, Bulgaria
- CHU, Clermont-Ferrand, France
- Hospital, Vigo, Spain
- Erciyes Üniversitesi Tıp Fakültesi, Kayseri, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 157 screened patients disposed as: 135 patients treated and randomised, 20 patients not included (reasons: screen failures: 14, protocol violation: 1, consent withdrawal: 4 and other reasons: 1) and 2 patients treated but not randomised.
Groups:
- T4020: 1 drop every other day during 5 days
  T4020
- Saline Solution: 1 drop every other day during 5 days
  Placebo
Period: Overall Study
Arm/Group | T4020 | Saline Solution
Started | 71 | 64
Completed | 71 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T4020 | Saline Solution | Total
Number analyzed (Participants) | 71 | 64 | 135
Age, Categorical [Count of Participants; unit: Participants] — Population: 73 treated patients with T4020 but 2 patients treated but not randomised. These 2 patients were excluded from the mITT set.
  Participants
    <=18 years | 3 | 5 | 8
    Between 18 and 65 years | 68 | 59 | 127
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 73 treated patients with T4020 but 2 patients treated but not randomised. These 2 patients were excluded from the mITT set.
  years | 27.5 (7.9) | 28.9 (10.2) | 28.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 73 treated patients with T4020 but 2 patients treated but not randomised. These 2 patients were excluded from the mITT set.
  Participants
    Female | 21 | 20 | 41
    Male | 50 | 44 | 94
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: 73 treated patients with T4020 but 2 patients treated but not randomised. These 2 patients were excluded from the mITT set.
  participants
    Turkey | 19 | 18 | 37
    France | 21 | 17 | 38
    Bulgaria | 15 | 14 | 29
    Spain | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Healing of Corneal Epithelial Defect at Day 3
Time Frame: Day 3
Population: mITT set (135 participants) analysed results. 137 treated participants: 73 treated patients with T4020 but 2 patients treated but not randomised. These 2 patients were excluded from the mITT set.
Measure: Count of Participants; unit: Participants
Arm/Group | T4020 | Saline Solution
Number analyzed (Participants) | 71 | 64
Participants | 20 | 25

2. Primary Outcome: Number of Participants With Complete Healing of Corneal Epithelial Defect at Day 4
Time Frame: Day 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | T4020 | Saline Solution
Number analyzed (Participants) | 71 | 64
Participants | 47 | 47

3. Secondary Outcome: Corneal Epithelial Defect Size Assessment
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | T4020 | Saline Solution
Number analyzed (Participants) | 71 | 64
mm^2 | 1.0 (4.6) | 1.9 (6.9)

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Time Frame: Through study completion, an average of 1 month
Population: Safety set (137 treated participants)
Measure: Count of Participants; unit: Participants
Arm/Group | T4020 | Saline Solution
Number analyzed (Participants) | 73 | 64
Participants | 12 | 8

ADVERSE EVENTS:
Time Frame: From the first visit to the final visit performed by the patient + 1 month later, assessed up to 95 days
Description: Safety set: 137 participants. 137 treated participants: 73 treated patients withT4020 but 2 patients treated but not randomised. These 2 patients were excluded from the mITT set.mITT set (135 participants) analysed results.
Arm/Group | T4020 | Saline Solution
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/64
Other Adverse Events (participants affected / at risk) | 12/73 | 8/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T4020 (N=73) | Saline Solution (N=64)
Conjunctival hyperaemia (Eye disorders) | 3 (3) | 1 (1) — Ocular adverse event
Malabsorption from application site (General disorders) | 1 (1) | 0 (0) — Ocular adverse events
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) — Ocular adverse event
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Systemic Non Ocular adverse event
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) — Systemic Non Ocular adverse event
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Systemic Non Ocular adverse event
Headache (Nervous system disorders) | 3 (3) | 0 (0) — Systemic Non Ocular adverse event
Contact lens intolerance (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event
Corneal disorder (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event
Corneal infiltrates (Eye disorders) | 0 (0) | 1 (1) — Ocular adverse event
Corneal oedema (Eye disorders) | 3 (3) | 2 (2) — Ocular adverse event
Corneal opacity (Eye disorders) | 2 (2) | 0 (0) — Ocular adverse event
Eye pain (Eye disorders) | 3 (3) | 1 (1) — Ocular adverse event
Eyelid oedema (Eye disorders) | 2 (2) | 0 (0) — Ocular adverse event
Keratitis (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2) — Ocular adverse event
Punctate keratitis (Eye disorders) | 2 (2) | 1 (1) — Ocular adverse event
Vision blurred (Eye disorders) | 1 (1) | 0 (0) — Ocular adverse event
Eye infection (Infections and infestations) | 1 (1) | 0 (0) — Ocular adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever form without prior written agreement of THEA.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT02979054/Prot_SAP_000.pdf